CLINICAL TRIAL: NCT06454227
Title: Antiseptic Washing Prior to Skin Closure During Cesarean Delivery- a Randomized Control Trial
Brief Title: Subcutaneous Lavage in Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: WASHCD-HMO-CTIL
Record Dates: First submitted 2024-05-07; First posted 2024-06-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-05

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subcutan lavage (Active Comparator): Subcutaneous washing with antiseptic solution: Chlorhexidine gluconate 0.2%
  Interventions: Procedure: Subcutaneous washing
- no lavage (Placebo Comparator): No subcutaneous washing
  Interventions: Procedure: no subcutaneous washing

INTERVENTIONS:
Procedure: Subcutaneous washing — subcutaneous washing with chlorhexidine gluconate prior to skin closure
  Arms: Subcutan lavage
Procedure: no subcutaneous washing — no washing
  Arms: no lavage

SUMMARY:
The goal of this clinical trial is to learn if antiseptic washing prior to skin closure during cesarean section reduces rates of surgical site infection.

intraoperative washing is a common practice in other surgical fields and several studies have shown efficacy in reducing postoperative infection rates. no randomized control trial has tested this intervention during cesarean section.

The main questions we aim to answer are:

Does subcutaneous antiseptic washing reduce the rates of surgical site infection? Does antiseptic washing improve scar healing? Does antiseptic washing reduce hospital stay, postpartum fever rates and readmission cases?

Researchers will compare subcutaneous antiseptic washing to no intervention to see if surgical site infection rates reduce

Participants will:

consent to participate in the trial Visit the postpartum clinic 30 days after surgery

ELIGIBILITY:
Inclusion Criteria:

* pregnant women undergoing cesarean delivery

Exclusion Criteria:

* pregnant women undergoing vaginal delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women undergoing cesarean delivery
Enrollment: 600 (Estimated)
Dates: Start 2024-09-22 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
surgical site infection | 30 days after surgery
  SSI infection rates

SECONDARY OUTCOMES:
hospital stay | 30 days after surgery
  length of hospital stay
wound healing | 30 days after surgery
  assessment of the healing according to Southampton criteria: presence of inflammation, erythema or discharge
postpartum fever | 30 days after surgery
  fever recording

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No